CLINICAL TRIAL: NCT02225821
Title: Antibiotic Prophylaxis to Prevent Wound Infections Following Implant Removal
Brief Title: Wound Infections Following Implant Removal
Acronym: WIFI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); AO Research Fund (Other)
Responsible Party: Principal Investigator, J.C. Goslings, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SB155014; NTR 4393 (Other: Nederlands Trial Register)
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Surgical Wound Infection
Keywords: Implant Removal; Antibiotic Prophylaxis; Postoperative wound infection; Orthopedics
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antibiotic prophylaxis (Active Comparator): a single gift of 1000 mg cefazolin in 10 cc of NaCl 0.9% (intervention group)
  Interventions: Drug: Cephalozin
- No antibiotic prophylaxis (Placebo Comparator): a single gift of 10 cc NaCl 0.9%, given in the same manner (control group).
  Interventions: Other: Sodium chloride

INTERVENTIONS:
Drug: Cephalozin — 1000 mg Cephalozin
  Other Names: Kefzol
  Arms: antibiotic prophylaxis
Other: Sodium chloride — 10 cc of NaCl 0.9%
  Other Names: NaCl 0.9%
  Arms: No antibiotic prophylaxis

SUMMARY:
In the Netherlands about 18,000 surgical procedures with implant removal are annually performed after fracture healing, of which 30-80% concern the foot, ankle and lower leg region. For clean surgical procedures, the rate of postoperative wound infections (POWIs) should be less than 5%. However, rates of 10-12% following implant removal, specifically after foot, ankle and lower leg fractures are reported. Currently, surgeons decide individually if antibiotics prophylaxis is given, since no guideline exists. This leads to undesirable practice variation.

Therefore, the investigators propose a double-blind randomized controlled trial (RCT) in patients scheduled for implant removal following a foot, ankle or lower leg fracture, to assess the (cost-)effectiveness of a single gift of antibiotic prophylaxis. Primary outcome is a POWI within 30 days after implant removal. Secondary outcomes are quality of life, functional outcome at 30 days and 6 months after implant removal and costs.

With 2 x 250 patients a decrease in POWI from 10% to 3.3% (expected rate in clean-contaminated elective orthopedic trauma procedures) can be detected (Power=80%, 2-sided alpha=5%, including 15% lost to follow up).

If the assumption of the investigators, that prophylactic antibiotics prior to implant removal reduces the infectious complication rate, is confirmed by this RCT, this will offer a strong argument to adopt a single gift of antibiotic prophylaxis as standard practice of care. This will reduce the incidence of POWIs and consequently will lead to less physical and social disabilities and health care use. In addition, it will decrease the rate of use of empiric broad-spectrum antibiotics (and antibiotic resistance) prescribed upon suspicion or diagnosis of a POWI. A preliminary, conservative estimation suggests yearly cost savings in the Netherlands of €3.5 million per year.

DETAILED DESCRIPTION:
See study protocol

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years and ≤75 years of all ethnic backgrounds
* Implant removal following foot, ankle and/or lower leg surgery

Exclusion Criteria:

* Removing and re-implanting osteosynthesis material in the same session
* Active wound infection or (plate) fistula
* Antibiotic treatment at time of elective implant removal for a concomitant disease or infection
* A medical history of an allergic reaction to a cephalosporin, penicillin, or any other β-lactam antibiotic.
* Insufficient comprehension of the Dutch language to understand the patient information to make an informed decision to participate.
* Kidney disease (eGFR <60 ml/min/1.73m^2).
* Treatment with probenecide, anticoagulants (see SPC)
* Pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Postoperative wound infection (POWI) | 30 days
  The primary outcome variable is a POWI within 30 days after implant removal as defined by the criteria applied by the Centers for Disease and Control.

SECONDARY OUTCOMES:
Health-related quality of life | baseline, one month, 6 months
  Health-related quality of life (as measured by the EQ-5D questionnaire)
Functional outcome | baseline, 1 month, 6 months
  Functional outcome following implant removal as assessed with the Lower Extremity Functional Scale (LEFS). The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention
Patient satisfaction | 1 month, 6 months
  Patient satisfaction following implant removal as measured by a ten-point Visual Analog Scale
Health care resources utilization | baseline, 1 month, 6 months
  Health care resources utilization at baseline, 1 month and 6 months after implant removal (including amongst others, number of visits to the general practitioner and use of home care organizations) as measured by way of a combination of the Dutch iMTA Medical Consumption Questionnaire (iMCQ) and iMTA Productivity Cost Questionnaire (iPCQ) (adapted to the study setting).

OTHER OUTCOMES:
Costs | Costs per quality adjusted life year
  Costs (economic evaluation including budget impact analysis): the economic evaluation of antibiotic prophylaxis in patients scheduled for implant removal (following a foot, ankle or lower leg fracture) against no prophylaxis as its best alternative will be performed as a cost-effectiveness (CEA) as well as a cost-utility (CUA) analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Manouk Backes, MD, MSc, Study Chair — Academic Medical Center/Sint Lucas Andreas Hospital; Tim Schepers, MD, PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (21):
- Netherlands (21):
  - Medisch Centrum Alkmaar, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Amstelland Ziekenhuis, Amstelveen
  - Academic Medical Center, Amsterdam
  - BovenIJ Ziekenhuis, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Sint Lucas Andreas Ziekenhuis, Amsterdam
  - VU Medisch Centrum, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf, Delft
  - Deventer Ziekenhuis, Deventer
  - Catharina Ziekenhuis, Eindhoven
  - Elkerliek Ziekenhuis, Helmond
  - Tergooiziekenhuizen, Hilversum
  - Spaarne Ziekenhuis, Hoofddorp
  - Westfries Gasthuis, Hoorn
  - Rijnland Ziekenhuis, Leiderdorp
  - Vlietland Ziekenhuis, Schiedam
  - MC Haaglanden, The Hague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Backes M, Schep NW, Luitse JS, Goslings JC, Schepers T. Indications for implant removal following intra-articular calcaneal fractures and subsequent complications. Foot Ankle Int. 2013 Nov;34(11):1521-5. doi: 10.1177/1071100713502466. Epub 2013 Sep 13. PMID 24038057
- [Background] Backes M, Dingemans SA, Schep NW, Bloemers FW, Van Dijkman B, Garssen FP, Haverlag R, Hoogendoorn JM, Joosse P, Mirck B, Postma V, Ritchie E, Roerdink WH, Sintenie JB, Soesman NM, Sosef NL, Twigt BA, Van Veen RN, Van der Veen AH, Van Velde R, Vos DI, De Vries MR, Winkelhagen J, Goslings JC, Schepers T. Wound Infections Following Implant removal below the knee: the effect of antibiotic prophylaxis; the WIFI-trial, a multi-centre randomized controlled trial. BMC Surg. 2015 Feb 6;15:12. doi: 10.1186/1471-2482-15-12. PMID 25972101
- [Derived] Backes M, Dingemans SA, Dijkgraaf MGW, van den Berg HR, van Dijkman B, Hoogendoorn JM, Joosse P, Ritchie ED, Roerdink WH, Schots JPM, Sosef NL, Spijkerman IJB, Twigt BA, van der Veen AH, van Veen RN, Vermeulen J, Vos DI, Winkelhagen J, Goslings JC, Schepers T; WIFI Collaboration Group. Effect of Antibiotic Prophylaxis on Surgical Site Infections Following Removal of Orthopedic Implants Used for Treatment of Foot, Ankle, and Lower Leg Fractures: A Randomized Clinical Trial. JAMA. 2017 Dec 26;318(24):2438-2445. doi: 10.1001/jama.2017.19343. PMID 29279933